CLINICAL TRIAL: NCT06810492
Title: A Single-arm Exploratory Study of the Efficacy and Safety of CDK4/6 Inhibitors in Combination with Endocrine Therapy in the Neoadjuvant Treatment of HR+/HER2- Early Breast Cancer
Brief Title: The Efficacy and Safety of CDK4/6 Inhibitors in Combination with Endocrine Therapy in the Neoadjuvant Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hongmei Zheng, PhD (Other)
Responsible Party: Sponsor-Investigator, Hongmei Zheng, PhD, director, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBCHBCC011
Record Dates: First submitted 2024-12-30; First posted 2025-02-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Stage III; Breast Cancer Stage II
Keywords: Hormone receptor (HR) positive; HER2 negative; neoadjuvant treatment; CDK4/6 inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; abemaciclib; palbociclib; dalpiciclib; Letrozole; Anastrozole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HR+/HER2- breast cancer patients who are intolerance or insensitivity to neoadjuvant chemotherapy (Experimental): 1. Age ≥ 18 years old.
  2. Premenopausal and postmenopausal stage II-III females or males (patients with multicenter and/or multifocal early-invasive breast cancer) if all histopathological examination of tumors meet the pathological criteria of ER and/or PR>10% and HER2- (HER2 expression 0 or 1+ or 2+ and negative FISH test).
  3. Intolerance or insensitivity to neoadjuvant chemotherapy: 2 cycles of neoadjuvant chemotherapy, tumor evaluation PD/SD, advanced age, and inability to tolerate chemotherapy with underlying diseases.
  4. ECOG PS score 0-2
  Interventions: Drug: Ribociclib; abemaciclib; palbociclib; Dalpiciclib

INTERVENTIONS:
Drug: Ribociclib; abemaciclib; palbociclib; Dalpiciclib — Neoadjuvant therapy: CDK4/6 inhibitor combined with endocrine, a total of 6 cycles, 1 cycle every 28 days.
  CDK4/6 inhibitors (choose one of the following four types):
  * Dalpiciclib 125 mg orally once a day d1-21 every 28 days for a cycle (3 weeks/1 week off)
  * Palbociclib 125 mg orally once a day, d1-21, every 28 days in cycles (3 weeks/1 week off)
  * Abemaciclib 150 mg orally twice daily in 28-day cycles (may be reduced to 100 mg orally twice daily if not tolerated)
  * Ribociclib 400 mg orally once a day in a 28-day cycle Endocrine therapy drugs: take according to the label. Premenopausal patients need to be treated for ovarian function suppression.
  Other Names: Letrozole; Anastrozole; Esomeprazole

SUMMARY:
To explore the efficacy and safety of CDK4/6 inhibitors combined with endocrine neoadjuvant therapy for stage II-III HR-positive/HER2-negative breast cancer.

This study adopts a single-arm, open-label design, and plans to include 40 patients with stage II-III HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Premenopausal and postmenopausal stage II-III females or males (patients with multicenter and/or multifocal early-invasive breast cancer) if all histopathological examination of tumors meet the pathological criteria of ER and/or PR>10% and HER2- (HER2 expression 0 or 1+ or 2+ and negative FISH test).
3. Patients must have histologically confirmed ER and/or PR >10%, HER2-, early invasive breast cancer.
4. Intolerance or insensitivity to neoadjuvant chemotherapy: 2 cycles of neoadjuvant chemotherapy, tumor evaluation PD/SD, advanced age, and inability to tolerate chemotherapy with underlying diseases.
5. ECOG PS score 0-2.
6. Patients must be able and willing to swallow and retain oral medications.
7. Premenopausal women within 14 days of enrollment, or women with amenorrhea for less than 12 months at the time of enrollment, must have a negative serum or urine pregnancy test.
8. Patients who have received neoadjuvant endocrine therapy are eligible for enrollment as long as they are enrolled within 6 months of initial histologic diagnosis and have completed no more than 2 months of neoadjuvant endocrine therapy.
9. Absolute neutrophil count ≥ 1500/µL, platelet ≥ 100000/mm3, hemoglobin ≥ 10g/dL

Exclusion Criteria:

1. Prior treatment with any CDK inhibitor.
2. Inflammatory breast cancer or stage IV breast cancer or bilateral breast cancer.
3. History of anaphylaxis caused by chemical or biologic components similar to dalsily.
4. Patients who have received any drugs or substances with effective CYP3A isoenzyme inhibitors or inducers within 7 days of enrollment.
5. Uncontrolled intercurrent illness that would limit compliance with study requirements.
6. Pregnant women or women of childbearing potential with a negative pregnancy test within 14 days prior to admission.
7. Patients with any history of malignancy are not eligible.
8. Patients who have received endocrine therapy within 5 years prior to the diagnosis of the current malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At the end of Cycle 6 (each cycle is 28 days)
  The main effect evaluation index was Objective response rate (ORR) after CDK4/6 inhibitor combined with endocrine, a total of 6 cycles.

SECONDARY OUTCOMES:
Ki67 variations | At the end of Cycle 2(each cycle is 28 days)
  Tumor samples were collected by surgical resection during the screening period (mandatory), at the time of treatment for 8 weeks (mandatory), and at the time of surgery (mandatory). Each test center was responsible for collecting samples, and the Hubei cancer Hospital determined the levels of Ki67.
complete cell cycle arrest (CCCA; Ki67 ≤ 2.7%) | 6 months
  Ki67 levels were assessed through serial biopsies at baseline , before ET treatment and C2D28 after ET treatment
iDFS | 2 years
  Disease free survival for 3 years and 5 years, which means the rate of patients without local recurrence and distant metastasis in the whole patients at the same group will be calculated with Kaplan Meier survival curves.
QoL | 1 year
  Life quality score was evaluated by European Organization of Research and treatment of Cancer-Questionnaire of Life Quality-C30 Version 3 (EORTC-QLQ-C30 V3), which conduct a series of questions about the patients' physical condition, activity of daily life, adverse reaction and mood condition. The range in the questionnaire for the score is from 1 to 4, in which 1 stands for having no discomfort and 4 stands for having great discomfort.

IPD SHARING:
Plan to Share IPD: Yes
Baseline data of enrolled patients, endocrine therapeutics, and idfs